CLINICAL TRIAL: NCT03750695
Title: Acute Effects of Aerobic and Resistance Exercise on Maternal Glucose Metabolism and Vascular Function in Obese Pregnancy
Brief Title: Acute Exercise Effects in Obese Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105627
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-05

CONDITIONS: Pregnancy Complications; Obesity; Pre-Eclampsia; Gestational Diabetes
Keywords: exercise; glucose; vascular
MeSH Terms: conditions — Pregnancy Complications; Obesity; Pre-Eclampsia; Diabetes, Gestational; Motor Activity | interventions — Resistance Training; Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Single group crossover design of acute effects of resistance exercise, aerobic exercise or rest (control) on maternal vascular function and glucose metabolism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute Resistance Exercise (Experimental): One acute exercise session of 40 minutes of resistance exercise
  Interventions: Behavioral: Resistance exercise
- Acute Aerobic Exercise (Experimental): One acute session of 40 minutes of aerobic exercise
  Interventions: Behavioral: Aerobic Exercise
- Acute Resting Session (Placebo Comparator): One session of 40 minutes of quiet rest
  Interventions: Behavioral: Rest

INTERVENTIONS:
Behavioral: Resistance exercise — One acute exercise session of resistance exercise (40 minutes including 3 sets of 8-10 repetitions at the participant's 10 repetition maximum load of upper and lower extremity exercise
  Arms: Acute Resistance Exercise
Behavioral: Aerobic Exercise — One acute session of aerobic exercise (40 minutes of cycle ergometry exercise at 70% of VO2peak)
  Arms: Acute Aerobic Exercise
Behavioral: Rest — 40 minutes of quiet rest in semi-recumbent position
  Arms: Acute Resting Session

SUMMARY:
Obesity before and during pregnancy is associated with a higher risk for a number of obstetric and metabolic complications in women and their offspring. Of particular importance, obese women have a higher risk of developing gestational diabetes and preeclampsia. In addition, obese women have larger offspring who have a higher risk for the development of obesity and diabetes; both largely attributed to higher maternal glycemia and glucose intolerance during pregnancy. Thus, identifying rehabilitative interventions that improve maternal and offspring metabolic and cardiovascular health in obese pregnancy are critical and have immediate and generational impact. Resistance and aerobic exercise training is a clinical staple for improving musculoskeletal, metabolic and cardiovascular health in non-gravid adolescents and adults with obesity however little is known regarding the effects of exercise during obese pregnancy. This study proposes to collect preliminary data on the independent effects of acute aerobic and resistance rehabilitative exercise on glucose metabolism and vascular function during pregnancy in n=15 obese women in order to inform a large, multisite clinical trial examining the acute and chronic effects of aerobic and resistance exercise on glucose metabolism and vascular function in normal weight, overweight and obese women during pregnancy.

DETAILED DESCRIPTION:
Maternal obesity prevalence is at a historic high with over 1 in 3 women entering pregnancy obese and 1 in 10 extremely obese. Obesity before and during pregnancy is associated with a higher risk for a number of obstetric and metabolic complications in women and their offspring. Of particular importance, obese women have a higher risk of developing gestational diabetes and preeclampsia. In addition, obese women have larger offspring who have a higher risk for the development of obesity and diabetes; both largely attributed to higher maternal glycemia and glucose intolerance during pregnancy. Thus, identifying rehabilitative interventions that improve maternal and offspring metabolic and cardiovascular health in obese pregnancy are critical and have immediate and generational impact.

Resistance and aerobic exercise training is a clinical staple for improving musculoskeletal, metabolic and cardiovascular health in non-gravid adolescents and adults with obesity. Observational studies suggest that exercise in pregnancy is safe and higher levels of physical activity before and during pregnancy in normal weight (i.e. lean) women reduces the risk of gestational diabetes and gestational hypertensive disorders; however, little is known regarding the effects of exercise training during obese pregnancy and several important questions still exist. These include: 1) "What are the acute and chronic effects of maternal exercise on glucose metabolism and vascular function?", 2) "Are there different effects of aerobic and resistance type exercise on glucose metabolism and vascular function?" and 3) "What are the physiologic and molecular transducers of maternal aerobic and resistance exercise for changes in maternal glucose metabolism and vascular function during pregnancy?" This pilot project aims to collect preliminary data on these questions.

This proposal would be the first study to collect preliminary data on the independent effects of acute aerobic and resistance rehabilitative exercise in pregnancy, and further, in obese women; a population with a high morbidity during gestation. In addition, this proposal would inform a large, multisite clinical trial examining the acute and chronic effects of aerobic and resistance exercise on glucose metabolism and vascular function in normal weight, overweight and obese women during pregnancy. Moreover, this proposal would provide initial evidence of molecular transducers of acute physical activity/rehabilitative exercise necessary for a large, comprehensive clinical trial examining the molecular transducers of rehabilitative exercise in normal weight, overweight and obese women during different stages of pregnancy.

Specific Aim #1: To characterize the acute effects of aerobic and resistance exercise on glucose metabolism (tolerance, insulin sensitivity and β-cell function) in obese women during mid-pregnancy.

Specific Aim #2: To characterize the acute effects of aerobic and resistance exercise on vascular function in obese women during mid-pregnancy.

Specific Aim #3: To explore the molecular transducers of physiologic responses in glucose metabolism and vascular function following acute aerobic and resistance exercise in obese women during mid-pregnancy.

The hypothesis is that acute aerobic and resistance rehabilitative exercise will improve post-exercise glucose metabolism and vascular function in obese women during mid-pregnancy. In a subsequent multi-site clinical trial, this study will examine differences in physiologic effects and molecular transducers of aerobic and resistance exercise on glucose metabolism and vascular function during different stages of pregnancy in overweight and obese women.

ELIGIBILITY:
Inclusion Criteria:

1. First trimester BMI ≥ 30.0 and <45.0 kg/m2 (calculated from clinical weight and height)
2. Singleton gestation, between 23 weeks and 0/7 days and 28 weeks and 0/7 days
3. Normal fetal anatomy (no major structural abnormalities identified on standard of care survey before enrollment)
4. Established prenatal care at Women's Health Clinic before 18 weeks of gestation, plans to deliver at Barnes-Jewish Hospital
5. Permission from Obstetrics physician provider to participate in study.

Exclusion Criteria:

1. Gestational or pre-gestational diabetes diagnosis
2. Inability to provide voluntary consent
3. Currently using illegal drugs (e.g., cocaine, methamphetamine, opiates) (safety risk and potential confounding)
4. Current smoker who does not agree to stop (confounding)
5. Participation in routine (>1x/week) exercise program (may improve glucose metabolism/vascular function)
6. History of heart disease, orthopedic, metabolic or neurological condition that would contraindicate exercise (safety risk)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Cade, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 3 interventions were: 1) 1-hour of rest, 2) 1-hour of resistance exercise, and 3) 1-hour of aerobic exercise. Each of these interventions were separated by 1-week. N=8 participants were randomized into performing these interventions in the order of rest-aerobic-resistance and n=8 participants in the order of rest-resistance-aerobic.
Groups:
- Rest, Then Aerobic Exercise, and Then Resistance Exercise Order: Rest: 40 minutes of quiet rest in semi-recumbent position
  Aerobic Exercise: One acute session of aerobic exercise (40 minutes of cycle ergometry exercise at 70% of VO2peak)
  Resistance exercise: One acute exercise session of resistance exercise (40 minutes including 3 sets of 8-10 repetitions at the participant's 10 repetition maximum load of upper and lower extremity exercise
  Participant performed interventions in order of rest, then aerobic exercise, then resistance exercise.
- Rest-Resistance-Aerobic Order: Rest: 40 minutes of quiet rest in semi-recumbent position Resistance exercise: One acute exercise session of resistance exercise (40 minutes including 3 sets of 8-10 repetitions at the participant's 10 repetition maximum load of upper and lower extremity exercise
  Aerobic Exercise: One acute session of aerobic exercise (40 minutes of cycle ergometry exercise at 70% of VO2peak)
  Participant performed interventions in order of rest, then resistance exercise, then aerobic exercise.
Period: Overall Study
Arm/Group | Rest, Then Aerobic Exercise, and Then Resistance Exercise Order | Rest-Resistance-Aerobic Order
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study. All participants were randomized to receive all interventions.
Groups:
- All Study Participants: Resistance exercise: One acute exercise session of resistance exercise (40 minutes including 3 sets of 8-10 repetitions at the participant's 10 repetition maximum load of upper and lower extremity exercise
  Aerobic Exercise: One acute session of aerobic exercise (40 minutes of cycle ergometry exercise at 70% of VO2peak)
  Rest: 40 minutes of quiet rest in semi-recumbent position
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Oral Glucose Insulin Sensitivity (OGIS) Index
Description: Oral Glucose Insulin Sensitivity (OGIS) during a 2-hour oral glucose tolerance test. OGIS (an acronym for Oral Glucose Insulin Sensitivity) is a method for the assessment of insulin sensitivity from the oral glucose tolerance test. OGIS provides an index which is analogous to the index of insulin sensitivity obtained from the glucose clamp. Mari, et al. OGIS uses modeling of glucose values at 0, 90, 120 min and insulin values at 0 and 90 min (2-h OGTT) to calculate the index. A model-based method for assessing insulin sensitivity from the oral glucose tolerance test. Diabetes Care 2001 Mar;24(3):539-48. The formula for OGIS is the following: (glucose clearance rate + square root(glucose clearance rate*glucose clearance rate + 4*pp5*pp6(glucose at 90 min-gcl)*330))/2. A calculation spreadsheet for OGIS is found at: http://webmet.pd.cnr.it/ogis/index.php
Time Frame: 2 hours post-intervention, up to approximately 3 hours
Population: Participants completed all interventions but in different order
Measure: Mean (Standard Deviation); unit: uU/mL
Groups:
- Acute Rest: 1-hour of sitting rest
Arm/Group | Acute Aerobic Exercise | Acute Resistance Exercise | Acute Rest
Number analyzed (Participants) | 15 | 15 | 15
uU/mL | 405.0 (56.9) | 426.0 (53.9) | 418.9 (67.0)

2. Primary Outcome: Percent Change in Endothelial Function
Description: Augmentation index: reactive hyperemic response post-blood pressure cuff inflation. Reactive hyperemia is the transient increase in organ blood flow that occurs following a brief period of ischemia (e.g., arterial occlusion).
Time Frame: baseline and immediately post-intervention, approximately 40 minutes
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Acute Rest: One session of 40 minutes of quiet rest
  Rest: 40 minutes of quiet rest in semi-recumbent position
Arm/Group | Acute Resistance Exercise | Acute Aerobic Exercise | Acute Rest
Number analyzed (Participants) | 15 | 15 | 15
percent change | 19.2 (11.0) | 20.3 (8.0) | 16.1 (7.7)
Statistical Analysis 1: Comparison: Acute Resistance Exercise vs Acute Aerobic Exercise vs Acute Rest; Repeated measures linear regression; Test type: Other; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: Approximately 3 hours after each intervention.
Arm/Group | Acute Resistance Exercise | Acute Aerobic Exercise | Acute Resting Session
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03750695/Prot_SAP_000.pdf